CLINICAL TRIAL: NCT01989104
Title: Cadence and Intensity in Children and Adolescents (CADENCE-KIDS)
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PBRC 13019; 1R21HD073807-01A1 (NIH)
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Results first posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: Indirect calorimetry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Children: 6-12 years of age
- Adolescents: 13-17 years of age
- Young adults: 18-20 years of age

SUMMARY:
The purpose of this study is to measure and link cadence (number of steps taken in a minute) to intensity of physical activity (e.g., low-intensity, moderate-intensity, vigorous-intensity) in children and adolescents (6-20 years-old), and to identify the cadence values corresponding to children's and adolescent's behavior during simulated free-living activities.

DETAILED DESCRIPTION:
Procedure - 1 visit - (approximately 3 hours in total)

Day of Testing: Participant must be FASTED - No food for 4 hours before visit. All of the study procedures involving the participant will be completed in a single testing session (one-day - approximately 3 hours) at the Pennington Biomedical Research Center. If preferred, two visits on separate days can be scheduled to complete the protocol.

* Screening questions (approximately 3-5 minutes)

  o Participants (or their legal guardian) will be asked to answer several screening questions to determine their eligibility for participating in CADENCE-KIDS.
* Height and weight measures data collection (approximately 10 minutes)

  * Height will be measured.
  * Body weight and body fat percentage will be measured using a specialized scale.
  * Waist circumference will then be measured using a measuring tape.
* Instrument attachment, treadmill walking, free-living activities (approximately 140 minutes)

  * Participants will be fitted with 10 devices (Digi-Walker Pedometer, NL-1000 Pedometer, StepWatch Activity Monitor, SenseWear Armband, GT3X+ accelerometer, GENEActiv Accelerometer, Actical Accelerometer, ActivPal Accelerometer, Polar Heart Rate Monitor, K4b2 Portable Metabolic Unit) to measure/monitor physical activity throughout the testing session.
  * Participants will then complete several low intensity free-living activities while their physical activity and oxygen uptake are concurrently assessed. Specifically, participants will rest in a chair, watch a portion of a child-friendly movie while seated in a chair, and color in a coloring book while seated in a chair. Each activity will last for 5 minutes and a 2 minute rest will occur between each activity.
  * Participants will then complete a series of walking bouts on a treadmill while their physical activity and oxygen uptake are concurrently assessed. The walking bouts start at 0.5 miles per hour and end at 5 miles per hour (0.5 miles per hour increments). Treadmill testing stops when the participant finishes the bout where they naturally select to jog/run, or following the completion of the last bout at 5.0 miles per hour, whichever occurs first. A 2 minute rest will occur between each treadmill bout.
  * Participants will then complete three additional free-living activities where physical activity and oxygen uptake continue to be concurrently measured. Specifically, participants will step up and down on an aerobic step at 88 beats per minute, dribble a basketball, and perform jumping jacks at 126 beats per minute (63 jumping jacks per minute). Each activity will last for 5 minutes and a 2 minute rest will occur between each activity.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 20 years of age at the time of study enrollment
* Not limited in the ability to walk

Exclusion Criteria:

* Hospitalization for mental illness within the past 5 years.
* Any condition/medication that may affect heart rate response to exercise testing.
* Previous history of, or clinical symptoms or signs of, cardiovascular disease, stroke or transient ischemic attacks, chest pain, unusual dyspnea during physical activity/exercise, severe ankle edema, or intermittent claudication.
* Previous history of musculoskeletal injuries or problems causing severe pain during physical activity or exercise which interferes with daily activities.
* Participant has a pacemaker or other implanted medical device (including metal joint replacements).
* Participant is pregnant.
* Participant is unable to complete all testing (1 or two sessions, as preferred) within a maximal two week period.

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2013-12; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catrine Tudor-Locke, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Gould ZR, Mora-Gonzalez J, Aguiar EJ, Schuna JM Jr, Barreira TV, Moore CC, Staudenmayer J, Tudor-Locke C. A catalog of validity indices for step counting wearable technologies during treadmill walking: the CADENCE-Kids study. Int J Behav Nutr Phys Act. 2021 Jul 16;18(1):97. doi: 10.1186/s12966-021-01167-y. PMID 34271922
- [Derived] Tudor-Locke C, Schuna JM Jr, Han H, Aguiar EJ, Larrivee S, Hsia DS, Ducharme SW, Barreira TV, Johnson WD. Cadence (steps/min) and intensity during ambulation in 6-20 year olds: the CADENCE-kids study. Int J Behav Nutr Phys Act. 2018 Feb 26;15(1):20. doi: 10.1186/s12966-018-0651-y. PMID 29482554

RESULTS

PARTICIPANT FLOW:
Groups:
- Children Group 1: 6-8 years of age
- Children Group 2: 9-11 years of age
- Adolescents Group 1: 12-14 years of age
- Adolescents Group 2: 15-17 years of age
Period: Overall Study
Arm/Group | Children Group 1 | Children Group 2 | Adolescents Group 1 | Adolescents Group 2 | Young Adults
Started | 25 | 25 | 25 | 24 | 24
Completed | 22 | 25 | 25 | 24 | 24
Not Completed | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Children Group 1 | Children Group 2 | Adolescents Group 1 | Adolescents Group 2 | Young Adults | Total
Number analyzed (Participants) | 22 | 25 | 25 | 24 | 24 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 25 | 25 | 24 | 0 | 96
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 24 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 13 | 12 | 12 | 60
  Male | 12 | 12 | 12 | 12 | 12 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 5 | 10 | 11 | 7 | 42
  White | 11 | 19 | 15 | 13 | 17 | 75
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 25 | 25 | 24 | 24 | 120

OUTCOME MEASURES:

1. Primary Outcome: Cadence - Steps Per Minute
Description: Cadence steps per minute represents an overlooked opportunity to describe the intensity of ambulatory activity.
Time Frame: 1 day
Measure: Mean (99% Confidence Interval); unit: Cadence - Steps per Minute
Arm/Group | Children Group 1 | Children Group 2 | Adolescents Group 1 | Adolescents Group 2 | Young Adults
Number analyzed (Participants) | 22 | 25 | 25 | 24 | 24
Cadence - Steps per Minute
  Moderate Intensity | 128.4 [121.7 to 134.5] | 116.5 [109.3 to 123.9] | 106.6 [102.5 to 111.0] | 101.3 [97.5 to 104.8] | 87.3 [79.4 to 95.7]
  Vigorous Intensity | 157.7 [151.8 to 164.0] | 142.7 [134.6 to 152.8] | 129.3 [124.1 to 135.6] | 126.3 [122.9 to 129.8] | 129.9 [126.3 to 133.6]

ADVERSE EVENTS:
Time Frame: 8 hours
Description: 0 affected
Arm/Group | Children Group 1 | Children Group 2 | Adolescents Group 1 | Adolescents Group 2 | Young Adults
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/25 | 0/25 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/25 | 0/25 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/22 | 0/25 | 0/25 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT01989104/Prot_SAP_000.pdf